CLINICAL TRIAL: NCT01535521
Title: Evaluation of Sleep Position Trainer for Positional Sleep Apnea Patients After Therapy With Mandibular Advancement Device (MAD)
Brief Title: Sleep Positional Trainer for Positional Sleep Apnea After Mandibular Advancement Device (MAD) Therapy
Acronym: SupPos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethisch Comité UZ Antwerpen (Other)
Responsible Party: Sponsor-Investigator, Ethisch Comité UZ Antwerpen, Dr. Olivier M. Vanderveken (principal investigator), University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Other Study IDs: SupPos
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Positional Sleep Apnea; Mandibular Advancement Device

ARMS (1):
- SPT in patients with MAD (Other)
  Interventions: Device: Sleep Position Trainer (SPT)

INTERVENTIONS:
Device: Sleep Position Trainer (SPT)

SUMMARY:
The investigators will perform a clinical trial comparing mandibular advancement device (MAD) therapy with sleep positional trainer (SPT) and the combination of MAD and SPT in patients with positional sleep apnea using MAD. Patients are invited for 2 consecutive polysomnographies (PSGs) in randomized order: one PSG with SPT, one PSG with SPT and MAD. PSGs are performed at the Antwerp University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients with supine dependent Obstructive Sleep Apnea (OSA) after Mandibular Advancement Device (MAD) Therapy: Apnea Hypopnea Index (AHI) supine ≥ 2x AHI non supine
* 5 < AHI < 50/h sleep on polysomnography (PSG) with MAD in situ
* ≥ 20% supine position during PSG with the MAD in situ
* AHI non-supine < 10/h en AHI supine ≥ 10/h on PSG with MAD in situ
* Unchanged Body Mass Index (BMI)(BMI ± 1 kg/m²) at moment of inclusion compared to BMI at baseline PSG

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Dieltjens M, Vroegop AV, Verbruggen AE, Wouters K, Willemen M, De Backer WA, Verbraecken JA, Van de Heyning PH, Braem MJ, de Vries N, Vanderveken OM. A promising concept of combination therapy for positional obstructive sleep apnea. Sleep Breath. 2015 May;19(2):637-44. doi: 10.1007/s11325-014-1068-8. Epub 2014 Oct 22. PMID 25335642